CLINICAL TRIAL: NCT04504331
Title: A Phase 1B Study of Infigratinib in Combination With Tamoxifen in Hormone Receptor Positive, HER2 Negative, FGFR Altered Advanced Breast Cancer
Brief Title: Study of Infigratinib in Combination With Tamoxifen in Hormone Receptor Positive, HER2 Negative, FGFR Altered Advanced Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug manufacturer decision to terminate development.
Sponsor: Jennifer Lee Caswell-Jin (Other)
Collaborators: National Cancer Institute (NCI) (NIH); QED Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Lee Caswell-Jin, Assistant Professor of Medicine (Oncology), Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-53650; BRS0113 (Other: OnCore); K08CA252457 (NIH); NCI-2020-13784 (Other: Clinical Trials Reporting Program)
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Results first posted 2023-06-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; HER2-negative Breast Cancer; ER Positive Breast Cancer; PR-Positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — infigratinib; Tamoxifen; Iohexol; Iopamidol; Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1: Infigratinib (100mg) + Tamoxifen (Experimental): In study part 1 (dose exploration), participants will receive up to infigratinib 100 mg. 100 mg of Infigratinib will be administered orally daily, 3 weeks on, 1 week off + 20 mg/day tamoxifen
  Interventions: Drug: Infigratinib; Drug: Tamoxifen; Drug: Omnipaque 350; Drug: Iopamidol; Diagnostic Test: Computed tomography (CT)
- Cohort 2: Infigratinib (125mg) + Tamoxifen (Experimental): In study part 1 (dose exploration), participants will receive up to infigratinib 125 mg. 125 mg of Infigratinib will be administered orally daily, 3 weeks on, 1 week off + 20 mg/ day tamoxifen
  Interventions: Drug: Infigratinib; Drug: Tamoxifen; Drug: Omnipaque 350; Drug: Iopamidol; Diagnostic Test: Computed tomography (CT)
- Cohort 3: Infigratinib (75mg) + Tamoxifen (Experimental): In study part 1 (dose exploration), participants will receive up to infigratinib 75 mg. 75 mg of Infigratinib will be administered orally daily, 3 weeks on, 1 week off + 20 mg/day tamoxifen
  Interventions: Drug: Infigratinib; Drug: Tamoxifen; Drug: Omnipaque 350; Drug: Iopamidol; Diagnostic Test: Computed tomography (CT)

INTERVENTIONS:
Drug: Infigratinib — Oral dose
  Other Names: FGFR 1-3-Selective Tyrosine Kinase Inhibitor; 872511-34-7; NVP-BGJ398; BGJ-398
Drug: Tamoxifen — Oral Dose
  Other Names: Nolvadex; Soltamox; Apo-Tamox; Tamofen; Tamone; ICI-46474
Drug: Omnipaque 350 — IV contrast agent
  Other Names: Iohexol; Hexopaque; Nycodenz; Exypaque; Compound 545
Drug: Iopamidol — IV contrast agent
  Other Names: Isovue 300; Isovue 370; Iopamiro; Iopamiron; Scanlux; Niopam; Jopamidol; Solutrast
Diagnostic Test: Computed tomography (CT) — Computed tomography (CT) to assess disease state using Iopamidol and/or Omnipaque 350.

SUMMARY:
The purpose of the study is identify the dose(s) of infigratinib to use in combination with tamoxifen to treat patients with a particular type of advanced breast cancer (hormone receptor-positive, HER2-negative, FGFR-altered breast cancer)

DETAILED DESCRIPTION:
Primary Objective: Determine the maximum (no greater than 125 mg) dose of infigratinib used in combination with the FDA-approved dose and schedule of tamoxifen (Cohort 1) in terms of the number of dose-limiting toxicities observed in the first 2 cycles of therapy in subjects with hormone receptor-positive, HER2-negative advanced breast cancer.

Secondary Objective:

* Estimate the incidence of treatment-emergent adverse events (serious and non-serious).
* Estimate the objective tumor response rate (ORR) in subjects with measurable disease.
* Estimate the progression-free survival (PFS).
* Estimate the durable clinical benefit rate.

ELIGIBILITY:
Inclusion Criteria:

* History of biopsy proven ER positive and/or PR positive, HER2 negative breast cancer and radiographic evidence of metastatic disease, or locally recurrent unresectable disease. ER positivity and PR positivity are defined as ≥ 1% cells staining positive by immunohistochemistry. HER2 negativity is defined by immunohistochemistry (IHC) or Fluorescence in situ hybridization (FISH).
* Cancer subtype: Predicted integrative subtype classification of IC2 or IC6 according classifier on targeted sequencing data from FoundationOne.
* Evaluable or measurable disease, by cohort. Cohort 1 only: Evaluable or measurable disease, as defined by RECIST v1.1. Bone only disease is acceptable.

Cohort 2 only: Measurable disease, as defined by RECIST v1.1.

* ≥ 18 years old
* Eastern Cooperative Oncology Group (ECOG) 0 to 2
* Prior cancer therapy (except for endocrine therapy, denosumab, or bisphosphonates) must be discontinued for 2 weeks prior to initiation of study drugs. Recovery from adverse events of previous cancer therapies to baseline or Grade 1 except for alopecia or stable Grade 2 neuropathy. Radiotherapy must also be completed at least 2 weeks prior to initiation of study drugs
* Absolute neutrophil count (ANC) ≥ 1,000/mm3
* Platelets ≥ 75,000/mm3
* Hemoglobin ≥ 9.0 g/dL
* Total bilirubin ≤ 1.8 mg/dL (unless documented Gilbert's disease)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 90 U/L
* Estimated glomerular filtration rate (GFR) ≥ 45 mL/min
* Phosphorus between 2.5 and 4.5 mg/dL, inclusive
* Total corrected (for albumin) serum calcium between 8.5 and 10.5 mg/dL, inclusive
* Amylase < 200 U/L
* Lipase < 120 U/L
* Ability to understand and the willingness to sign a written informed consent document
* Agrees to take sevelamer, if indicated, and has no contraindications to use of this medication (that is: known hypersensitivity to sevelamer or component of the formulation; bowel obstruction; active bowel mucosal injury such as ulcerative colitis or gastrointestinal bleeding).
* Agrees to follow low phosphate diet, if indicated
* Able to swallow and retain oral medication
* Women must be postmenopausal, defined as (at least one of):

  * ≥ 60 years of age;
  * amenorrhea for at least 24 months;
  * amenorrhea for at least 12 months with serum estradiol < 20 pg/mL;
  * prior bilateral oophorectomy; OR
  * treatment with a luteinizing hormone (LH) releasing hormone agonist (such as goserelin acetate or leuprolide acetate) initiated at least 28 days prior to study enrollment.
* Women being treated with a LH releasing agonist but who are otherwise of childbearing potential (did not undergo total hysterectomy or bilateral tubal ligation at least 6 weeks before first dose of study drug) must have a negative pregnancy test within 7 days of the first dose of study drug.
* Women who are being treated with a LH releasing agonist but are otherwise of childbearing potential must agree to use barrier contraception or an intrauterine device while taking study drug and for 3 months following their last dose of study drug. Alternatively, total abstinence is acceptable if preferred by the subject.
* Sexually active men must agree to use a condom during intercourse while taking drug and for 3 months after the last dose of the study drug and should not father a child during this period. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner to prevent delivery of the drug via seminal fluid.

Exclusion Criteria:

* History of another primary malignancy within 3 years except adequately treated in situ carcinoma of the cervix or non melanoma carcinoma of the skin or any other curatively treated malignancy that is not expected to require treatment for recurrence during the course of the study.
* Neurologic symptoms related to central nervous system metastases requiring increasing doses of corticosteroids. Note that subjects with central nervous system metastases are eligible if they are on a stable corticosteroid dose for at least 2 weeks preceding study entry.
* Current evidence of corneal or retinal disorder/keratopathy including, but not limited to, bullous/band keratopathy, corneal abrasion, inflammation/ulceration, keratoconjunctivitis, confirmed by ophthalmologic examination. Subjects with asymptomatic ophthalmologic conditions assessed by the investigator to pose minimal risk for study participation may be enrolled in the study.
* Current evidence of extensive tissue calcification including, but not limited to, the soft tissue, kidneys, intestine, myocardium, and lung with the exception of calcified lymph nodes, minor pulmonary parenchymal calcifications, and asymptomatic coronary calcification.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral infigratinib (eg, ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection).
* Current evidence of endocrine alterations of calcium/phosphate homeostasis, eg, parathyroid disorders, history of parathyroidectomy, tumor lysis, or tumoral calcinosis.
* Currently receiving or planning during study participation to receive treatment with agents that are known strong inducers or inhibitors of CYP3A4 and medications which increase serum phosphorus and/or calcium concentration. Subjects are not permitted to receive enzyme inducing anti epileptic drugs, including carbamazepine, phenytoin, phenobarbital, and primidone. See Appendix B for a list of prohibited concomitant medications and supplements.
* Has consumed grapefruit, grapefruit juice, grapefruit hybrids, pomegranates, star fruits, pomelos, Seville oranges, or products containing juice of these fruits within 7 days prior to first dose of study drug.
* Have used amiodarone within 90 days prior to first dose of study drug.
* Has used medications known to prolong the QT interval and/or are associated with a risk of Torsades de Pointes (TdP) 7 days prior to first dose of study drug. See Appendix B for a list of prohibited concomitant medications and supplements.
* Has used calcium or vitamin D within 3 days prior to first dose of study drug. Calcium supplementation may subsequently be used as clinically indicated (for hypocalcemia) on study.
* Have clinically significant cardiac disease including any of the following:

  1. Congestive heart failure requiring treatment (New York Heart Association Grade ≥ 2), left ventricular ejection fraction (LVEF) < 50% or local lower limit of normal as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO), or uncontrolled hypertension (refer to the European Society of Cardiology and European Society of Hypertension guidelines [Williams et al., 2018])
  2. Presence of Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grade ≥ 2 ventricular arrhythmias, atrial fibrillation, bradycardia, or conduction abnormality
  3. Unstable angina pectoris or acute myocardial infarction ≤ 3 months prior to first dose of study drug
  4. Corrected QT interval Fredericia (QTcF) > 470 msec (males and females). Note: If the QTcF is > 470 msec in the first electrocardiogram (ECG), a total of 3 ECGs separated by at least 5 minutes should be performed. If the average of these 3 consecutive results for QTcF is ≤ 470 msec, the subject meets eligibility in this regard.
  5. Known history of congenital long QT syndrome
* Have had a recent (≤ 3 months) transient ischemic attack or stroke.
* Pregnant or nursing woman.

  * All subject files must include supporting documentation to confirm subject eligibility. The method of confirmation can include, but is not limited to, laboratory test results, radiology test results, subject self report, and medical record review.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Lee Caswell-Jin, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was closed before any participants were enrolled in Cohort 3 (Infigratinib (75 mg) + Tamoxifen).
Groups:
- Cohort 1: Infigratinib (100mg) + Tamoxifen: In study part 1 (dose exploration), participants receive infigratinib up to 100 mg administered orally daily, 3 weeks on, 1 week off + 20 mg/day tamoxifen
- Cohort 2: Infigratinib (125mg) + Tamoxifen: In study part 1 (dose exploration), participants receive infigratinib up to 125 mg administered orally daily, 3 weeks on, 1 week off + 20 mg/ day tamoxifen
- Cohort 3: Infigratinib (75mg) + Tamoxifen: In study part 1 (dose exploration), participants receive infigratinib up to 75 mg administered orally daily, 3 weeks on, 1 week off + 20 mg/day tamoxifen
Period: Dose Level 1 (up to 18 28-day Cycles+FU)
Arm/Group | Cohort 1: Infigratinib (100mg) + Tamoxifen | Cohort 2: Infigratinib (125mg) + Tamoxifen | Cohort 3: Infigratinib (75mg) + Tamoxifen
Started | 3 | 0 | 0
Completed at Least 6 Treatment Cycles | 3 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Dose Level 2 (up to 18 28-day Cycles+FU)
Arm/Group | Cohort 1: Infigratinib (100mg) + Tamoxifen | Cohort 2: Infigratinib (125mg) + Tamoxifen | Cohort 3: Infigratinib (75mg) + Tamoxifen
Started | 0 | 1 | 0
Completed at Least 6 Treatment Cycles | 0 | 0 | 0
Completed | 0 | 1 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Infigratinib (100mg) + Tamoxifen | Cohort 2: Infigratinib (125mg) + Tamoxifen | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 1 | 0 | 1
Age, Continuous [Median (Standard Deviation); unit: years] | 55.2 (9.6) | 38.5 (NA) — Not calculable for a single value | 53.9 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose-limiting Toxicities (DLTs)
Description: The primary outcome for this study is dose-limiting toxicities (DLTs) during the first 2 cycles of therapy. All grades per the Common Terminology Criteria for Adverse Events (CTCAE). DLT is defined as a related and clinically significant adverse event (AE), including missed doses due to a related AE.
Time Frame: 8 weeks
Measure: Number; unit: DLTs
Arm/Group | Cohort 1: Infigratinib (100mg) + Tamoxifen | Cohort 2: Infigratinib (125mg) + Tamoxifen
Number analyzed (Participants) | 3 | 1
DLTs | 0 | 0

2. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAE)
Description: Treatment emergent adverse events (TEAEs) are defined as adverse events of any grade with initial onset or increasing in severity after the first dose of study treatment until 30 days after last dose of study drug. Pregnancy during the reporting period will be classified as a serious adverse event.
Time Frame: From first dose to 30 days after the last dose of study drug (up to 94 days)
Measure: Number; unit: adverse events
Arm/Group | Cohort 1: Infigratinib (100mg) + Tamoxifen | Cohort 2: Infigratinib (125mg) + Tamoxifen
Number analyzed (Participants) | 3 | 1
adverse events | 49 | 26

3. Secondary Outcome: Objective Tumor Response Rate
Description: Objective tumor response will be assessed as achieving a Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Complete Response (CR) or a Partial Response (PR). The outcome will be reported as the number of subjects that achieve an overall response (OR) to treatment, ie, CR or PR, within 18 months of starting treatment. RECIST criteria are:
  * CR = Disappearance of all target lesions
  * PR = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Overall Response (OR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s)
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
Time Frame: From enrollment to day of scan (up to 64 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Infigratinib (100mg) + Tamoxifen | Cohort 2: Infigratinib (125mg) + Tamoxifen
Number analyzed (Participants) | 3 | 1
Participants
  CR | 0 | 0
  PR | 0 | 0
  OR (CR + PR) | 0 | 0
  PD | 3 | 0
  SD | 0 | 1

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression free survival (PFS) means the participant remains alive without return or relapse of the tumor. The outcome is defined as the number of days to either progressive disease as defined per RECIST v1.1 or death. RECIST criteria are:
  * CR = Disappearance of all target lesions
  * PR = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Overall Response (OR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s)
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
Time Frame: up to 9 months
Measure: Median (Standard Deviation); unit: days
Arm/Group | Cohort 1: Infigratinib (100mg) + Tamoxifen | Cohort 2: Infigratinib (125mg) + Tamoxifen
Number analyzed (Participants) | 3 | 1
days | 61 (5.3) | NA — Not evaluable due to insufficient number of events

5. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit (CB) is defined as achieving a Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Complete Response (CR) ; Partial Response (PR); or Stable Disease (SD). The outcome will be reported as the number of subjects that achieve CR, PR, or SD. RECIST criteria are:
  * CR = Disappearance of all target lesions
  * PR = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * SD = Small changes that do not meet any of the above criteria
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s)
Time Frame: 6 months
Population: Participants who completed at least 6 treatment cycles are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Infigratinib (100mg) + Tamoxifen | Cohort 2: Infigratinib (125mg) + Tamoxifen
Number analyzed (Participants) | 3 | 0
Participants
  CR | 0 |
  PR | 0 |
  SD | 0 |
  CB (CR + PR +SD) | 0 |
  PD | 3 |

ADVERSE EVENTS:
Time Frame: Up to 9 months
Arm/Group | Cohort 1: Infigratinib (100mg) + Tamoxifen | Cohort 2: Infigratinib (125mg) + Tamoxifen
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Infigratinib (100mg) + Tamoxifen (N=3) | Cohort 2: Infigratinib (125mg) + Tamoxifen (N=1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) — Grade 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Infigratinib (100mg) + Tamoxifen (N=3) | Cohort 2: Infigratinib (125mg) + Tamoxifen (N=1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 1 (2) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Other - corneal endothelial cell count decreased (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysgeusia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Flushing (General disorders) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (6) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (2)
Immune system disorder (Immune system disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (4) | 1 (3)
Hypophosphtaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Chills (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Contusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia of lower extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Muscular weakness (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Vision blurred (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Other - pulling sensation in uterus (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Other - yeast infection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Contusion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Other - Eyelash thickening (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Vascular disorders) | 1 (1) | 0 (0)
Contusion (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Retinopathy (Vascular disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT04504331/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT04504331/ICF_000.pdf